CLINICAL TRIAL: NCT05888961
Title: Single-center Prospective Longitudinal Study of Taste in Patients With Cognitive Disorders at Different Stages of Severity (Isolated Cognitive Complaint, Minor or Major Neurocognitive Alzheimer-type Disorders) by Analysis of Gustatory Evoked Potentials
Acronym: MAPEG 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: JACQUIN 2023
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Disorders
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Blood Specimen Collection; Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control subjects (Active Comparator)
  Interventions: Biological: Blood samples; Other: Interviewing the subject and scales; Other: Neurocognitive evaluation; Other: Taste tests; Other: Computerized food preference questionnaires; Other: Nutritional status - body composition
- Subjects with an isolated cognitive complaint (Experimental)
  Interventions: Biological: Blood samples; Other: Interviewing the subject and scales; Other: Neurocognitive evaluation; Other: Taste tests; Other: Computerized food preference questionnaires; Other: Nutritional status - body composition
- Subjects with minor neurocognitive disorders (Experimental)
  Interventions: Biological: Blood samples; Other: Interviewing the subject and scales; Other: Neurocognitive evaluation; Other: Taste tests; Other: Computerized food preference questionnaires; Other: Nutritional status - body composition
- Subjects with major neurocognitive disorders of the mild to moderate Alzheimer's disease type (Experimental)
  Interventions: Biological: Blood samples; Other: Interviewing the subject and scales; Other: Neurocognitive evaluation; Other: Taste tests; Other: Computerized food preference questionnaires; Other: Nutritional status - body composition

INTERVENTIONS:
Biological: Blood samples — Fasting at the first session for hormonal measurements of leptin, insulin, acylated and non-acylated ghrelin, serotonin, albumin, protidemia and blood glucose.
  Repeated at 6 and 12 months for follow-up
Other: Interviewing the subject and scales — Collection of sociodemographic data, personal and family neurological history, treatments, MADRS depression scale and CDR autonomy scale.
  Carried out at the 1st session
Other: Neurocognitive evaluation — cognitive complaint questionnaire (CCQ), taste, smell, MoCA and MMSE (if not performed in the previous 6 months) Carried out at the 1st session. Repeated at 6 and 12 months for follow-up.
Other: Taste tests — Sweet and salty flavors at the 1st session and acid and umami flavors at the 2nd session. Repeated at 6 and 12 months for follow-up.
  Placement of electrodes on the scalp, recording of gustatory evoked potentials, subjective gustatory evaluation by means of visual analogue scales rated from 0 to 10, identification and naming of each of the primary flavors
Other: Computerized food preference questionnaires — Performed at the 1st session on a tactile tablet. Repeated at 6 and 12 months for follow-up.
Other: Nutritional status - body composition — Measurement of anthropometric data, bioelectrical impedancemetry (measurement of fat mass, lean mass, water mass and bone mass in kg), measurement of blood pressure and heart rate Performed at the 2nd session Repeated at 6 and 12 months for follow-up.

SUMMARY:
The aim of the MAPEG 2 study is to explore gustatory function and to follow its evolution in the 4 following groups of participants:

* Healthy subjects
* Participants with isolated cognitive complaint
* Participants with minor neurocognitive disorder
* Participants with mild and moderate Alzheimer-type major neurocognitive disorders

For this purpose, we want to compare the results of the following tests:

* Subjective taste tests (tasting solutions, answering food preference questionnaires),
* Gustatory evoked potential (GEP) parameters, recorded by electrodes placed on the scalp,
* And nutritional parameters (hormones of food intake by blood test, measurement of the global body composition).

Identifying and following the evolution of early taste disorders in case of cognitive disorders could improve the diagnosis of Alzheimer's disease in two ways:

* To allow an early diagnosis of Alzheimer's disease, and thus improve its management,
* To define groups of subjects at risk of developing Alzheimer's disease in later years.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent.
* For patients with mild to moderate Alzheimer's disease, the primary caregiver and the patient will be asked to provide oral consent
* Person of legal age
* Body Mass Index (BMI) < 30 kg/m².
* For the healthy group: absence of cognitive complaints and normal neurological assessment
* Patients meeting the criteria for isolated cognitive complaint: presence of cognitive complaint but normal neuropsychological evaluation
* Patients meeting diagnostic criteria for minor cognitive impairment: imaging (brain MRI) and neuropsychological assessment with a Clinical Dementia Rating (CDR) score of 0.5
* Patients meeting diagnostic criteria for mild to moderate Alzheimer's disease: imaging (brain MRI), neuropsychobiological criteria (consultation with neuropsychological assessment, CSF biomarkers), MMSE score ≥ 20 and CDR score of 1 or 1.5
* Fasting for at least 2 hours before GEP measurement

Exclusion Criteria:

* MMSE score<15
* Known COVID-19 infection within 6 months prior to inclusion
* Person not affiliated to national health insurance system
* Person under a legal protection measure (curatorship, guardianship)
* Person subject to a measure of legal protection
* Pregnant, parturient or breastfeeding women
* Subjects with a pacemaker (contraindication to bioelectrical impedance measurement)
* Adult unable to express consent or to perform cognitive tests.
* Active smoker (> 4 cigarettes per day on a regular basis)
* Diabetic subject (type 1 or type 2)
* Subject with acute or chronic ENT disease
* Treatment interfering with gustation
* Brain MRI showing another cause of neurocognitive disorder (except for vascular lesions Fazekas 1 accepted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Amplitude of the gustatory evoked potentials | After a 2-hour fasting period
Gustatory evoked potentials latency | After a 2-hour fasting period

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France